CLINICAL TRIAL: NCT01524926
Title: Cross-tumoral Phase 2 Clinical Trial Exploring Crizotinib (PF-02341066) in Patients With Advanced Tumors Induced by Causal Alterations of ALK and/or MET ("CREATE")
Brief Title: CREATE: Cross-tumoral Phase 2 With Crizotinib
Acronym: CREATE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-90101; 2011-001988-52 (EudraCT Number)
Record Dates: First submitted 2012-01-24; First posted 2012-02-02 (Estimated); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Locally Advanced and/or Metastatic Anaplastic Large Cell Lymphoma; Locally Advanced and/or Metastatic Inflammatory Myofibroblastic Tumor; Locally Advanced and/or Metastatic Papillary Renal Cell Carcinoma Type 1; Locally Advanced and/or Metastatic Alveolar Soft Part Sarcoma; Locally Advanced and/or Metastatic Clear Cell Sarcoma; Locally Advanced and/or Metastatic Alveolar Rhabdomyosarcoma
Keywords: Phase 2; Crizotinib; Anaplastic large cell lymphoma; Inflammatory myofibroblastic tumor; Papillary renal cell carcinoma type 1; Alveolar soft part sarcoma; Clear cell sarcoma; Alveolar rhabdomyosarcoma
MeSH Terms: conditions — Lymphoma, Large-Cell, Anaplastic; Granuloma, Plasma Cell; Sarcoma, Alveolar Soft Part; Sarcoma, Clear Cell; Rhabdomyosarcoma, Alveolar | interventions — Crizotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Crizotinib in Anaplastic large cell lymphoma (Experimental)
  Interventions: Drug: Crizotinib (PF-02341066)
- Crizotinib in Inflammatory myofibroblastic tumor (Experimental)
  Interventions: Drug: Crizotinib (PF-02341066)
- Crizotinib in Papillary renal cell carcinoma type 1 (Experimental)
  Interventions: Drug: Crizotinib (PF-02341066)
- Crizotinib in Clear cell sarcoma (Experimental)
  Interventions: Drug: Crizotinib (PF-02341066)
- Crizotinib in Alveolar soft part sarcoma (Experimental)
  Interventions: Drug: Crizotinib (PF-02341066)
- Crizotinib in Alveolar rhabdomyosarcoma (Experimental)
  Interventions: Drug: Crizotinib (PF-02341066)

INTERVENTIONS:
Drug: Crizotinib (PF-02341066) — For patients of 15yo and older, Capsules of 200 and 250 mg Daily dose of 500, 400 or 250 mg/day depending on toxicitie; for patients younger than 15yo, 280 mg/m²/dose BID, with reductions allowed to 80% as first reduction and to 60% as second reduction respectively of the initial dose.

SUMMARY:
The study will primarily assess the antitumor activity of crizotinib in a variety of tumors with alterations in ALK and/or MET pathways. The targeted patient population will include patients with tumors harboring specific alterations leading to ALK and/or MET activation, where tyrosine kinase inhibitors against these targets have not yet been adequately explored.

ELIGIBILITY:
General inclusion criteria:

* Locally advanced and/or metastatic anaplastic large cell lymphoma
* Locally advanced and/or metastatic inflammatory myofibroblastic tumor
* Locally advanced and/or metastatic papillary renal cell carcinoma type 1
* Locally advanced and/or metastatic alveolar soft part sarcoma
* Locally advanced and/or metastatic clear cell sarcoma
* Locally advanced and/or metastatic alveolar rhabdomyosarcoma.
* The above malignancies must be incurable by conventional surgery, radiotherapy, systemic therapy or any other means.
* Proven presence of specific ALK and/or MET pathway alteration in tumor tissue is not mandatory for patient registration.
* Availability of tumor material for central pathology review
* Written informed consent
* Measurable disease according to RECIST 1.1
* Patients with brain metastases are eligible if treated and/or neurologically stable with no ongoing requirement for corticosteroids (off steroids for at least 2 weeks) and not taking contraindicated medications. Absence of spinal cord compression unless treated with the patient attaining good pain control and stable or recovered neurologic function.
* No carcinomatous meningitis or leptomeningeal disease.
* Any previous systemic anticancer therapy must have been completed at least 4 weeks prior to initiation of study medication.
* No treatment with any other investigational drug within the past 4 weeks or within less than 4 half-life times of the investigational drug before treatment with crizotinib (whatever is the longest period).
* No prior therapy directly targeting ALK and/or MET, no previous treatment with crizotinib.
* Major surgery must have been completed at least 4 weeks prior to initiation of study medication.
* Prior palliative radiotherapy must have been completed at least 24 hrs prior to initiation of study medication, and minor surgical procedures must have been completed at least two weeks prior to the initiation of study medication.
* Eastern Cooperative Oncology Group (ECOG) performance status 0-2, or Lansky play scale ≥ 50 for children aged 1 to 12 yo
* Adequate hematological function: ANC ≥ 1 x 109/L, platelets ≥ 30 x 109/L and hemoglobin ≥ 8 g/dL.
* Adequate bone marrow, renal and hepatic functions
* All related adverse events from previous therapies must have recovered to ≤ Grade 1 (except alopecia). No persistence of adverse events from prior anti-cancer therapy deemed clinically relevant.
* No acute or chronic severe gastrointestinal conditions such as diarrhea or ulcerations.
* Normal cardiac function and no cerebrovascular accident including transient ischemic attack.
* No current congestive heart failure.
* No ongoing cardiac dysrhythmias of NCI CTCAE Grade >2.
* No uncontrolled atrial fibrillation of any grade.
* QTc interval <470 msec.
* Absence of interstitial lung disease.
* No concurrent use of drugs or foods that are known strongCYP3A4 inhibitors
* No concurrent use of drugs that are known potent CYP3A4 inducers,within 12 days prior to first dose of crizotinib
* No concomitant intercurrent illnesses
* Effective contraception method (if applicable)

Disease-specific inclusion criteria for patients with anaplastic large cell lymphoma

* Patient may have received previous systemic treatment, surgery and/or radiotherapy for localized, locally advanced or advanced disease.
* Patient must have received previous systemic chemotherapy (usually a CHOP-like multidrug combination, if not medically contraindicated, with or without monoclonal antibodies), and may not qualify for further conventional therapy with curative intent.
* No pretreatment limitations (including autologous or allogeneic stem cell- or bone marrow transplantation), provided all other patient selection criteria are met.

Disease-specific inclusion criteria for patients with inflammatory myofibroblastic tumor

* Patient may have received previous systemic treatment, surgery and/or radiotherapy for localized, locally advanced or metastatic disease.
* No mandatory pretreatment.
* No pretreatment limitations, provided all other patient selection criteria are met.

Disease-specific inclusion criteria for patients with papillary renal cell carcinoma type 1

* Patient may have received previous systemic treatment, surgery and/or radiotherapy for localized, locally advanced or metastatic disease.
* No mandatory pretreatment.
* No pretreatment limitations, provided all other patient selection criteria are met.

Disease-specific inclusion criteria for patients with clear cell sarcoma

* Patient may have received previous systemic treatment, surgery and/or radiotherapy for localized, locally advanced or metastatic disease.
* No mandatory pretreatment.
* No pretreatment limitations, provided all other patient selection criteria are met.

Disease-specific inclusion criteria for patients with alveolar soft part sarcoma

* Patient may have received previous systemic treatment, surgery and/or radiotherapy for localized, locally advanced or metastatic disease.
* No mandatory pretreatment.
* No pretreatment limitations, provided all other patient selection criteria are met.

Disease-specific inclusion criteria for patients with alveolar rhabdomyosarcoma

* Patient may have received previous systemic treatment, surgery and/or radiotherapy for localized, locally advanced or metastatic disease.
* Patient must have received previous systemic chemotherapy (usually anthracycline-based, if not medically contraindicated), and may not qualify for further conventional therapy with curative intent.
* No pretreatment limitations, provided all other patient selection criteria are met.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 582 (Estimated)
Dates: Start 2012-09 (Actual); Primary Completion 2017-12-06 (Actual); Study Completion 2022-10-30 (Actual)

PRIMARY OUTCOMES:
Antitumor activity of crizotinib
  To study the antitumor activity of crizotinib across predefined tumor types in patients whose tumors are harboring specific alterations in ALK and/or MET

SECONDARY OUTCOMES:
Safety (reporting of adverse events according to CTCAE v4.0)
Progression free survival
Disease control rate
Overall survival
Duration of response
Correlative research endpoints

CONTACTS AND LOCATIONS:
Locations (25):
- Belgium (2):
  - Hôpitaux Universitaires Bordet-Erasme - Institut Jules Bordet, Brussels
  - U.Z. Gasthuisberg, Leuven
- France (5):
  - Institut Bergonie, Bordeaux
  - Centre Georges-Francois-Leclerc, Dijon
  - Centre Leon Berard, Lyon
  - Assistance Publique - Hôpitaux de Marseille - Hôpital de La Timone, Marseille
  - Institut Gustave Roussy, Villejuif
- Germany (6):
  - Helios Klinikum Bad Saarow, Bad Saarow
  - Universitaetsklinikum Carl Gustav Carus, Dresden
  - Universitaetsklinikum - Essen, Essen
  - Medizinische Hochschule Hannover, Hanover
  - UniversitaetsMedizin Mannheim, Mannheim
  - Klinikum Grosshadern Ludwig-Maximilians Univ. Muenchen, München
- Fondazione IRCCS Istituto Nazionale dei Tumori, Milan, Italy
- Netherlands (3):
  - Leiden University Medical Centre, Leiden
  - Radboud University Nijmegen Medical Centre, Nijmegen
  - Erasmus MC - Sophia kindersiekenhuis, Rotterdam
- Oslo University Hospital - Radiumhospitalet, Oslo, Norway
- Maria Sklodowska-Curie Memorial Cancer Centre, Warsaw, Poland
- National Cancer Institute, Bratislava, Slovakia
- The Institute Of Oncology, Ljubljana, Slovenia
- United Kingdom (4):
  - St. James's University Hospital, Leeds
  - University College Hospital, London
  - Christie NHS Foundation Trust, Manchester
  - Nottingham University Hospitals NHS Trust - City Hospital, Nottingham

REFERENCES:
- [Derived] Schoffski P, Kubickova M, Wozniak A, Blay JY, Strauss SJ, Stacchiotti S, Switaj T, Bucklein V, Leahy MG, Italiano A, Isambert N, Debiec-Rychter M, Sciot R, Lee CJ, Speetjens FM, Nzokirantevye A, Neven A, Kasper B. Long-term efficacy update of crizotinib in patients with advanced, inoperable inflammatory myofibroblastic tumour from EORTC trial 90101 CREATE. Eur J Cancer. 2021 Oct;156:12-23. doi: 10.1016/j.ejca.2021.07.016. Epub 2021 Aug 13. PMID 34392187
- [Derived] Schoffski P, Sufliarsky J, Gelderblom H, Blay JY, Strauss SJ, Stacchiotti S, Rutkowski P, Lindner LH, Leahy MG, Italiano A, Isambert N, Debiec-Rychter M, Sciot R, Van Cann T, Marreaud S, Nzokirantevye A, Collette S, Wozniak A. Crizotinib in patients with advanced, inoperable inflammatory myofibroblastic tumours with and without anaplastic lymphoma kinase gene alterations (European Organisation for Research and Treatment of Cancer 90101 CREATE): a multicentre, single-drug, prospective, non-randomised phase 2 trial. Lancet Respir Med. 2018 Jun;6(6):431-441. doi: 10.1016/S2213-2600(18)30116-4. Epub 2018 Apr 15. PMID 29669701
- [Derived] Schoffski P, Wozniak A, Leahy MG, Aamdal S, Rutkowski P, Bauer S, Richter S, Grunwald V, Debiec-Rychter M, Sciot R, Geoerger B, Marreaud S, Collette S, Nzokirantevye A, Strauss SJ. The tyrosine kinase inhibitor crizotinib does not have clinically meaningful activity in heavily pre-treated patients with advanced alveolar rhabdomyosarcoma with FOXO rearrangement: European Organisation for Research and Treatment of Cancer phase 2 trial 90101 'CREATE'. Eur J Cancer. 2018 May;94:156-167. doi: 10.1016/j.ejca.2018.02.011. Epub 2018 Mar 20. PMID 29567632
- [Derived] Schoffski P, Wozniak A, Kasper B, Aamdal S, Leahy MG, Rutkowski P, Bauer S, Gelderblom H, Italiano A, Lindner LH, Hennig I, Strauss S, Zakotnik B, Anthoney A, Albiges L, Blay JY, Reichardt P, Sufliarsky J, van der Graaf WTA, Debiec-Rychter M, Sciot R, Van Cann T, Marreaud S, Raveloarivahy T, Collette S, Stacchiotti S. Activity and safety of crizotinib in patients with alveolar soft part sarcoma with rearrangement of TFE3: European Organization for Research and Treatment of Cancer (EORTC) phase II trial 90101 'CREATE'. Ann Oncol. 2018 Mar 1;29(3):758-765. doi: 10.1093/annonc/mdx774. PMID 29216400
- [Derived] Schoffski P, Wozniak A, Stacchiotti S, Rutkowski P, Blay JY, Lindner LH, Strauss SJ, Anthoney A, Duffaud F, Richter S, Grunwald V, Leahy MG, Reichardt P, Sufliarsky J, van der Graaf WT, Sciot R, Debiec-Rychter M, van Cann T, Marreaud S, Lia M, Raveloarivahy T, Collette L, Bauer S. Activity and safety of crizotinib in patients with advanced clear-cell sarcoma with MET alterations: European Organization for Research and Treatment of Cancer phase II trial 90101 'CREATE'. Ann Oncol. 2017 Dec 1;28(12):3000-3008. doi: 10.1093/annonc/mdx527. PMID 28950372